CLINICAL TRIAL: NCT00408590
Title: Phase I Trial of Intraperitoneal Administration of a) a CEA-Expressing Derivative, and b) a NIS-Expressing Derivative Manufactured From a Genetically Engineered Strain of Measles Virus in Patients With Recurrent Ovarian Cancer
Brief Title: Recombinant Measles Virus Vaccine Therapy and Oncolytic Virus Therapy in Treating Patients With Progressive, Recurrent, or Refractory Ovarian Epithelial Cancer or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000515008; P30CA015083 (NIH); MC0117 (Other: Mayo Clinic Cancer Center); 1260-03 (Other: Mayo Clinic - IRB); NCI-2009-01199 (Registry Identifier: CTRP); P50CA136393 (NIH)
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: ovarian clear cell cystadenocarcinoma; ovarian endometrioid adenocarcinoma; primary peritoneal cavity cancer; ovarian mixed epithelial carcinoma; ovarian mucinous cystadenocarcinoma; ovarian serous cystadenocarcinoma; ovarian undifferentiated adenocarcinoma; recurrent ovarian epithelial cancer; Brenner tumor
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Brenner Tumor | interventions — Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental Arm (Experimental)
  Interventions: Biological: carcinoembryonic antigen-expressing measles virus; Biological: oncolytic measles virus encoding thyroidal sodium iodide symporter; Genetic: reverse transcriptase-polymerase chain reaction; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: carcinoembryonic antigen-expressing measles virus
Biological: oncolytic measles virus encoding thyroidal sodium iodide symporter
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: A gene-modified virus may be able to kill tumor cells without damaging normal cells.

PURPOSE: This phase I trial is studying the side effects and best dose of an attenuated oncolytic measles virus therapy and oncolytic virus therapy in treating patients with progressive, recurrent, or refractory ovarian epithelial cancer or primary peritoneal cancer (measles virus vaccine therapy study closed as of 06/02/2008).

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and toxicity of recombinant carcinoembryonic antigen (CEA)-expressing measles virus (MV-CEA) and oncolytic measles virus encoding thyroidal sodium iodide symporter (MV-NIS) in patients with progressive, recurrent, or refractory ovarian epithelial or primary peritoneal cavity cancer ( MV-CEA closed as of 06/02/2008).
* Determine the maximum-tolerated dose of MV-CEA and MV-NIS in these patients ( MV-CEA closed as of 06/02/2008).
* Characterize viral gene expression at each dose level as manifested by CEA titers in these patients.
* Assess viremia, viral replication, and measles virus shedding or persistence after study therapy.
* Determine humoral and cellular immune response to the injected virus in these patients.
* Assess, preliminarily, the antitumor efficacy of this therapy, by assessing CA-125 levels, radiographic response, and time to progression, in these patients.
* Determine the time course of viral gene expression and virus elimination and biodistribution of virally infected cells at various time points after infection with MV-NIS using single photon emission computed tomography (SPECT/CT) imaging.
* Assess viremia, viral replication, and measles virus shedding/persistence following intraperitoneal administration of MV-NIS.

OUTLINE: This is a dose-escalation study.

Patients receive recombinant carcinoembryonic antigen-expressing measles virus (MV-CEA) or oncolytic measles virus encoding thyroidal sodium iodide symporter (MV-NIS) intraperitoneally over 30 minutes on day 1. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity ( MV-CEA closed as of 06/02/2008).

Cohorts of 3-6 patients receive escalating doses of MV-CEA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity ( MV-CEA closed as of 06/02/2008).

Peripheral blood mononuclear cells are collected at baseline and periodically during and after treatment to assess viremia. Throat gargle and urine specimens are assessed periodically during course 1 for viral shedding by reverse transcriptase-polymerase chain reaction (RT-PCR). Peritoneal aspirate is tested at baseline and periodically during treatment for viral replication by RT-PCR, co-culture with Vero cells, and measles virus N-specific mRNA in situ hybridization.

Patients may undergo single photon emission computed tomography (SPECT/CT) imaging at baseline and periodically during study.

After completion of study therapy, patients are followed periodically for up to 15 years.

PROJECTED ACCRUAL: A total of 46 patients will be accrued for this study.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years.
* Must have persistent, recurrent or progressive ovarian cancer or primary peritoneal cancer after prior treatment with platinum and taxol compounds. Histologic confirmation of the original primary tumor is required. Prior bilateral oophorectomy is required.
* Patients with the following histologic epithelial cell types are eligible: Serous adenocarcinoma, endometroid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma NOS
* The following laboratory values obtained ≤7 days prior to registration:

  * ANC ≥ 1500/μL
  * PLT ≥ 100,000/μL
  * Total bilirubin ≤ upper normal limit
  * AST ≤ 2 x ULN
  * Creatinine ≤ 1.5 x ULN
  * Hgb ≥ 9.0 g/dL
* Ability to provide informed consent.
* Willingness to return to Mayo Clinic Rochester for follow-up.
* Life expectancy ≥ 12 weeks.
* Must have anti-measles immunity as demonstrated by serum IgG anti-measles antibody levels of ≥ 20.0 EU/ml as determined by Enzyme Immunoassay (Diamedix, FL).
* Must have normal serum CEA levels (<5 mg/ml) both at the time of study entry and in any prior testing. (NOTE: Not applicable for the MV-NIS cohort.)
* Willingness to provide all biologic specimens as required by the protocol.
* Measurable disease by exam or CT scan, or, for patients with CA-125 elevation or with microscopic residual but without measurable disease on imaging, willingness to undergo laparoscopy for evaluation of treatment effect if no radiographic progression after 6 treatment cycles.
* CD4 count ≥200/μL or ≥15% of peripheral blood lymphocytes

Exclusion criteria:

* Epithelial tumors of low malignant potential, stromal tumors, and germ cell tumors of the ovary.
* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy. Subjects will be excluded if this is their first relapse and they have recurred >6 mo from completion of primary (adjuvant) chemotherapy.
* ECOG performance status (PS) 3 or 4.
* Active infection ≤5 days prior to registration.
* History of tuberculosis or history of PPD positivity.
* History of other malignancy ≤5 years except for non-melanoma skin cancer or carcinoma in situ of the cervix.
* Any of the following prior therapies:

  * Chemotherapy ≤ 3 weeks prior to study entry
  * Immunotherapy ≤ 4 weeks prior to study entry
  * Biologic therapy ≤ 4 weeks prior to study entry
  * Extensive abdominal surgery if it includes enterotomy(ies) <3 weeks prior to study entry. This criterion does not apply to placement of the peritoneal port-a-cath or lysis of adhesions at the time of study entry.
  * Any viral or gene therapy prior to study entry
* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment.
* New York Heart Association classification III or IV, known symptomatic coronary artery disease, or symptoms of coronary artery disease on systems review, or known cardiac arrhythmias (atrial fibrillation or SVT).
* Requiring blood product support.
* CNS metastases or seizure disorder.
* HIV-positive test result, or history of other immunodeficiency.
* History of organ transplantation.
* History of chronic hepatitis B or C.
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-FDA-approved indication and in the context of a research investigation).
* Any concurrent medications which could interfere with the trial.
* Intra-abdominal disease > 8 cm in diameter at the time of registration, intrahepatic disease, or disease beyond the abdominal cavity.
* Treatment with oral/systemic corticosteroids, with the exception of topical or inhaled steroids.
* Exposure to household contacts ≤15 months old or household contact with known immunodeficiency.
* Allergy to measles vaccine or history of severe reaction to prior measles vaccination.
* Allergy to iodine. This does not include reactions to intravenous contrast materials.

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2004-04-19 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2017-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1, Dose Level 1: Cohort 1 consists of the first 21 patients accrued to the study before addendum13. At dose level 1, these patients received a 10^3 TCID50dose of MV-CEA diluted in 500 ml of normal saline over 30 minutes. They receive treatment every 4 weeks for a total of 6 cycles.
- Cohort 1, Dose Level 2: Cohort 1 consists of the first 21 patients accrued to the study before addendum13. At dose level 2, these patients received a 10^4 TCID50dose of MV-CEA diluted in 500 ml of normal saline over 30 minutes. They receive treatment every 4 weeks for a total of 6 cycles.
- Cohort 1, Dose Level 3: Cohort 1 consists of the first 21 patients accrued to the study before addendum13. At dose level 3, these patients received a 10^5 TCID50dose of MV-CEA diluted in 500 ml of normal saline over 30 minutes. They receive treatment every 4 weeks for a total of 6 cycles.
- Cohort 1, Dose Level 4: Cohort 1 consists of the first 21 patients accrued to the study before addendum13. At dose level 4, these patients received a 10^6 TCID50dose of MV-CEA diluted in 500 ml of normal saline over 30 minutes. They receive treatment every 4 weeks for a total of 6 cycles.
- Cohort 1, Dose Level 5: Cohort 1 consists of the first 21 patients accrued to the study before addendum13. At dose level 5, these patients received a 10^7 TCID50dose of MV-CEA diluted in 500 ml of normal saline over 30 minutes. They receive treatment every 4 weeks for a total of 6 cycles.
- Cohort 1, Dose Level 6: Cohort 1 consists of the first 21 patients accrued to the study before addendum13. At dose level 6, these patients received a 10^8 TCID50dose of MV-CEA diluted in 500 ml of normal saline over 30 minutes. They receive treatment every 4 weeks for a total of 6 cycles.
- Cohort 1, Dose Level 7: Cohort 1 consists of the first 21 patients accrued to the study before addendum13. At dose level 7, these patients received a 10^9 TCID50dose of MV-CEA diluted in 500 ml of normal saline over 30 minutes. They receive treatment every 4 weeks for a total of 6 cycles.
- Cohort 2, Dose Level 1: Cohort 2 consists of the last 16 patients accrued to the study after addendum13. At dose level 1, these patients received one 0.025mg tablet of Cytomel 3 times a day for the 7 days leading up to a 10^8 TCID50 treatment of MV-NIS(every 4 weeks for up to 6 cycles). After this main treatment, they also received 5 mCi of Iodine, orally on days 3 and 8.
- Cohort 2, Dose Level 2: Cohort 2 consists of the last 16 patients accrued to the study after addendum13. At dose level 2, these patients received one 0.025mg tablet of Cytomel 3 times a day for the 7 days leading up to a 10^9 TCID50 treatment of MV-NIS(every 4 weeks for up to 6 cycles). After this main treatment, they also received 5 mCi of Iodine, orally on days 3 and 8.
Period: Overall Study
Arm/Group | Cohort 1, Dose Level 1 | Cohort 1, Dose Level 2 | Cohort 1, Dose Level 3 | Cohort 1, Dose Level 4 | Cohort 1, Dose Level 5 | Cohort 1, Dose Level 6 | Cohort 1, Dose Level 7 | Cohort 2, Dose Level 1 | Cohort 2, Dose Level 2
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 13
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Includes all dose levels of Cohort 1
- Cohort 2: Includes all dose levels of Cohort 2
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 21 | 16 | 37
Age, Continuous [Median (Full Range); unit: years] | 57 [43 to 82] | 57.5 [35 to 82] | 57 [35 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 16 | 37
Ascites Present [Number; unit: participants with ascites] | 7 | 13 | 20

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity
Description: If one patient experiences a Dose limiting Toxicity(DLT), up to three additional patients will be treated at the same dose level. If DLT is observed in only one of six patients treated at a given dose level, the next cohort of three patients will be treated at the next higher dose level. If two or more patients experience DLT at a particular dose level, then the dose escalation will cease and any subsequent patients will be treated at a lower dose level. Thus finding the Max tolerated dose
Time Frame: up to 12 months after last treatment
Population: All patients that received study drug for at least 4 weeks were evaluated for dose limiting toxicities.
Measure: Number; unit: participants with DLTs
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 21 | 16
participants with DLTs | 0 | 0

2. Secondary Outcome: Number of Responses (Complete and Partial, Stable and Progressive Disease)
Description: Responses will be summarized separately for the MV-CEA virus and MV-NIS virus by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease. CA125 levels and time to progression will also be summarized descriptively. Modified Response Evaluation Criteria in Solid Tumors(RECIST v1.0) criteria will be used. For target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter(LD) of target lesions; Progression (PD): As least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD
Time Frame: up to 12 months after last treatment
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 21 | 16
participants
  CR | 0 | 0
  PR | 0 | 0
  SD | 14 | 13
  PD | 7 | 3

3. Secondary Outcome: Change in CA-125 Levels From Baseline to Last Recorded Value (up to 18 Months)
Description: CA-125 tests are measured in units per milliliter (U/mL) and taken every cycle (up to 6-28 day cycles) during treatment and every three months up to 12 months after treatment. The change in CA-125 is calculated as the baseline CA-125 value subtracted by the last recorded value of CA-125 (up to 18 months from baseline.
Time Frame: baseline and up to 18 months
Measure: Median (Full Range); unit: U/ml
Arm/Group | Cohort 1, Dose Level 1 | Cohort 1, Dose Level 2 | Cohort 1, Dose Level 3 | Cohort 1, Dose Level 4 | Cohort 1, Dose Level 5 | Cohort 1, Dose Level 6 | Cohort 1, Dose Level 7 | Cohort 2, Dose Level 1 | Cohort 2, Dose Level 2
Number analyzed (Participants) | 3 | 1 | 3 | 2 | 3 | 3 | 3 | 3 | 13
U/ml | -20.2 [-57 to 61] | 97 [97 to 97] | 52 [-26 to 4300] | 42.5 [-140 to 225] | 129 [4 to 216] | -112 [-261 to -5] | 11 [-8 to 21] | 1200 [6 to 2800] | 18 [-447 to 3033]

4. Secondary Outcome: Time to Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: up to 12 months after last treatment
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 21 | 16
Days | 55 [21 to 277] | 64.5 [26 to 277]

ADVERSE EVENTS:
Arm/Group | Cohort 1 | Cohort 2
Serious Adverse Events (participants affected / at risk) | 3/21 | 2/16
Other Adverse Events (participants affected / at risk) | 21/21 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=21) | Cohort 2 (N=16)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Peritoneal infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=21) | Cohort 2 (N=16)
Hemoglobin decreased (Blood and lymphatic system disorders) | 6 (8) | 6 (12)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (6) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (3) | 2 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Endocrine disorder (Endocrine disorders) | 0 (0) | 1 (1)
Extraocular muscle paresis (Eye disorders) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 6 (9) | 7 (10)
Abdominal pain (Gastrointestinal disorders) | 16 (36) | 16 (33)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (9) | 6 (11)
Diarrhea (Gastrointestinal disorders) | 11 (12) | 9 (15)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Flatulence (Gastrointestinal disorders) | 8 (13) | 7 (14)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (13) | 9 (13)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (6) | 8 (11)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 4 (9) | 9 (20)
Edema limbs (General disorders) | 5 (9) | 4 (4)
Fatigue (General disorders) | 13 (26) | 10 (24)
Fever (General disorders) | 10 (16) | 10 (22)
General symptom (General disorders) | 1 (1) | 2 (3)
Injection site reaction (General disorders) | 1 (2) | 0 (0)
Pain (General disorders) | 7 (17) | 4 (5)
Bladder infection (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (3) | 1 (4)
Alkaline phosphatase increased (Investigations) | 1 (1) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 2 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2)
Creatinine increased (Investigations) | 1 (1) | 2 (5)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (2)
Leukocyte count decreased (Investigations) | 1 (3) | 4 (9)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (5) | 3 (6)
Platelet count decreased (Investigations) | 0 (0) | 3 (6)
Serum cholesterol increased (Investigations) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 1 (4)
Weight loss (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 9 (14) | 3 (4)
Blood glucose increased (Metabolism and nutrition disorders) | 3 (7) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (11) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (9) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (11) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 3 (6)
Neurological disorder NOS (Nervous system disorders) | 2 (2) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 3 (7)
Speech disorder (Nervous system disorders) | 1 (1) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (3)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 2 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (5) | 3 (8)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes